CLINICAL TRIAL: NCT06299267
Title: The Effect of Dual Task on Manual Skill Performance in Children and Adolescents
Acronym: Dual-task
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Igdir University (Other)
Responsible Party: Principal Investigator, Sema Bugusan Oruc, Head of Physiotherapy and Rehabilitation Department, Igdir University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Igdir181
Record Dates: First submitted 2024-02-27; First posted 2024-03-07 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Child, Only; Adolescent Development
Keywords: children; adolescent; manual skill; dual-task

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- effect of dual task (Other): effect of dual task
  Interventions: Other: dual task conditions

INTERVENTIONS:
Other: dual task conditions — dual task conditions on manual skill tests

SUMMARY:
The aim of the study is to investigate the effect of dual-task conditions on manual dexterity performance in typically developing young people and children between the ages of 7-18.

MATERIAL AND METHOD:

* Demographic information, dominant extremity will be noted and the evaluation will begin by applying the Physical Activity Questionnaire for Children.
* The evaluations will primarily evaluate the child's performance on a single cognitive task
* The cognitive task will be the n-back task (counting down task) to be applied in accordance with the level of the child or adolescent.
* Using the Visual Analogue Scale (VAS), participants will be asked to score the difficulty of the cognitive task as a number between 0 and 10.
* the 9-Hole Test will be applied and the times will be recorded by asking to write a given paragraph.
* Dual task evaluations will be administered by giving a simultaneous cognitive task while administering the -9-Hole Test and writing a paragraph.
* In order to reveal the dual-task cost (DTC), dual-task performance will be subtracted from single-task performance and the difference will be calculated in seconds.

As a result of this study, manual dexterity performance and cognitive performance in single-task conditions in typically developing children and adolescents will be revealed. Additionally, changes in this performance will be detected in dual-task situations.

DETAILED DESCRIPTION:
In the literature, balance or walking postural tasks are mostly used in dual-task studies for typically developing children. However, dual task tasks performed during manual skills in daily life have not been adequately researched. The aim of the study is to investigate the effect of dual-task conditions on manual dexterity performance in typically developing young people and children between the ages of 7-18. Although studies on this subject are limited in the world, a comprehensive study is needed on children and young people in our country.

MATERIAL AND METHOD:

* Demographic information, dominant extremity will be noted and the evaluation will begin by applying the Physical Activity Questionnaire for Children.
* The evaluations will primarily evaluate the child's performance on a single cognitive task in a supported sitting position on a chair, without a motor task. The cognitive task will be the n-back task (counting down task) to be applied in accordance with the level of the child or young person.
* Using the Visual Analogue Scale (VAS), participants will be asked to score the difficulty of the cognitive task as a number between 0 and 10.
* In order to evaluate the single motor performance of manual skills, the 9-Hole Test will be applied and the times will be recorded by asking to write a given paragraph.
* Dual task evaluations will be administered by giving a simultaneous cognitive task while administering the 9-Hole Test and writing a paragraph.
* In order to reveal the dual-task cost (DTC), dual-task performance will be subtracted from single-task performance and the difference will be calculated in seconds.

As a result of this study, manual dexterity performance and cognitive performance in single-task conditions in typically developing children and adolescents will be revealed. Additionally, changes in this performance will be detected in dual-task situations.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 7-18,
* Not having a chronic disease.

Exclusion Criteria:

* Participants must have had a health problem or had an operation that would affect the musculoskeletal system or dexterity performance in the last year (EX: Distal radius fracture).
* Having concentration problems such as attention deficit hyperactivity disorder (ADHD).
* Not volunteering to participate in the study and not signing a consent form.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 77 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
single cognitive task | 1minute
  The cognitive task will be the n-back task (counting down task) to be applied in accordance with the level of the child or adolescent
Visual Analogue Scale (VAS) | 1minute
  Participants will be asked to score the difficulty of the cognitive task and motor task as a number between 0 and 10. High score indicates difficulty of the activity. (0= simple task; 10= difficult task almost Icannot do.)
9-Hole Peg Test.-Single task | 2minutes
  In order to evaluate the single motor performance of manual skills, the 9-Hole PegTest will be applied.
9-Hole Peg Test and writing a given paragraph.-Dual task | 2 minutes
  In order to evaluate the dual task performance the 9-Hole PegTest will be applied with a count-back task.
writing a given paragraph.-Single task | 3 minutes
  In order to evaluate the single motor performance of manual skills a paragraph will be written.
writing a given paragraph.-Dual task | 3 minutes
  In order to evaluate the dual task performance the paragraph will be written with a count-back task.

CONTACTS AND LOCATIONS:
Overall Officials: Sema Büğüşan Oruç, PhD, Principal Investigator — Igdir University
Locations (1):
- Iğdır University, Iğdır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wollesen B, Janssen TI, Muller H, Voelcker-Rehage C. Effects of cognitive-motor dual task training on cognitive and physical performance in healthy children and adolescents: A scoping review. Acta Psychol (Amst). 2022 Apr;224:103498. doi: 10.1016/j.actpsy.2022.103498. Epub 2022 Jan 25. PMID 35091209
- [Background] Rubsam M, Girolami GL, Bhatt T. Heterogeneity of Tasks and Outcome Measures in Dual Tasking Studies in Children With Cerebral Palsy: A Scoping Review. Phys Ther. 2024 Jan 1;104(1):pzad151. doi: 10.1093/ptj/pzad151. PMID 37941469
- [Background] Szturm T, Parmar ST, Mehta K, Shetty DR, Kanitkar A, Eskicioglu R, Gaonkar N. Game-Based Dual-Task Exercise Program for Children with Cerebral Palsy: Blending Balance, Visuomotor and Cognitive Training: Feasibility Randomized Control Trial. Sensors (Basel). 2022 Jan 19;22(3):761. doi: 10.3390/s22030761. PMID 35161508